CLINICAL TRIAL: NCT02926131
Title: Field Evaluation of a Point-Of-Care Test for Serum Bilirubin Levels in Infants Born in a Tropical Limited-resource Setting.
Brief Title: A Study to Evaluate a New Jaundice Stick Test
Acronym: Bilistick
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Shoklo Malaria Research Unit (Other)
Responsible Party: Sponsor
Other Study IDs: SMRU1606
Record Dates: First submitted 2016-09-22; First posted 2016-10-06 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-07

CONDITIONS: Jaundice; Serum Bilirubin
Keywords: stick test
MeSH Terms: conditions — Jaundice | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants: Infants requiring serum bilirubin (SBR) measurement seen in Wang Pha clinic (WPA) clinic.
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — * One full capillary tube (50µl blood) will be used to measure the Hct level and the routine SBR using the BR-501 bilirubin meter machine (non-study procedure).
  * An additional half- filled capillary tube (25µl blood) will be used for the SBR measurement with the Bilistick system

SUMMARY:
This is an observational prospective study. The main purpose is to evaluate the stability of the Bilistick system in a humid and hot climate compared to the quantitative test for serum bilirubin (SBR) measurement currently used, the BR-501 total bilirubin meter, kept in a controlled environment.

The secondary aim is to assess the operational feasibility of the Bilistick system in a tropical limited-resource setting, when used by locally trained nurses.

DETAILED DESCRIPTION:
Study procedure:

1. SBR will be measured in parallel with two tests during three distinct seasons. (Cold, hot, rainy). The Blood is from an extra capillary sample taken from a single heel prick done for routine SBR) BR-501 total bilirubin meter, the quantitative test for SBR currently used, will be kept in a controlled environment while the new bilirubin test (Bilistick system) will be exposed to tropical conditions.
2. Trained nurses will use the Bilistick system observed by a qualified laboratory technician; Usability of the Bilistick system by the trained nurses will be evaluated via a 5-point Likert scale questionnaire and focus groups discussions.

ELIGIBILITY:
Inclusion Criteria:

* Written or thumb print for informed consent from the parent
* Infant born ≥ 35 weeks of gestational age
* Infant who needs a routine SBR measurement
* Infant in stable clinical condition prior to SBR measurement confirmed by the trained nurses

Exclusion Criteria:

The participant will not be enrolled in the study if ANY of the following applies:

* Infant who already had 1 SBR measurement done with the Bilistick system
* Last haematocrit measurement > 65% or no previous haematocrit measurement

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infant seen in WPA clinic during the neonatal period (birth to 28 days of life).
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Comparison of the agreement of serum bilirubin measurement between the two tests in three different seasons | 18 months
  The main outcome of interest is the potential effect of environmental conditions on the quantitative outcome of the Bilistick System, using BR-501 bilirubin meter machine as a reference. The Bland-Altman analysis will be used to compare the two tests.
Within each season, evaluation of the impact of temporal variation on the agreement of serum bilirubin measurement between the two tests. | 18 months
  A linear regression analysis will be done to look for statistically significant effect of exposure time on the difference between the average total bilirubin serum levels of the two tests.

SECONDARY OUTCOMES:
Evaluation of the usability of the Bilistick system using a 5-point likert scale questionnaire and a focus group discussions | 18 months
  5-point likert scale questionnaire will be filled individually by the trained nurses at the end of each defined season. Quantitative variables related to the secondary outcomes will be measured with the mean, median and ratio according to the distribution of the variable and compared with appropriated statistical test.
Perception by the trained nurses of the Bilistick system usability with a focus group discussion (FGD). | 18 months
  The FGD will be centered around the answers obtained from the questionnaires and the concerns raised by the trained nurses and laboratory technicians during each recruitment period. Qualitative variable from the focus group will be analysed with Nvivo.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Rose McGready, MD, Principal Investigator — Shoklo Malaria Research Unit (SMRU)
Locations (1):
- Shoklo Malaria Research Unit (SMRU), Mae Sot, Changwat Tak, Thailand

IPD SHARING:
Plan to Share IPD: No